CLINICAL TRIAL: NCT03376321
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of Pimodivir in Combination With the Standard-of-Care Treatment in Adolescent, Adult, and Elderly Hospitalized Patients With Influenza A Infection
Brief Title: A Study to Evaluate the Efficacy and Safety of Pimodivir in Combination With the Standard-of-Care Treatment in Adolescent, Adult, and Elderly Hospitalized Participants With Influenza A Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated early (date of study termination decision: 28 August 2020) as a result of the outcome of the pre-planned Interim Analysis.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108399; 2017-002156-84 (EudraCT Number); 63623872FLZ3001 (Other: Janssen Research & Development, LLC)
Expanded Access: NCT03834376 (No longer available)
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Results first posted 2021-04-14 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Influenza A
MeSH Terms: interventions — pimodivir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm 1 (pimodivir + Standard-of-Care [SOC] treatment) (Experimental): Participants will receive pimodivir 600 milligram (mg) orally twice daily for 5 days (on Days 1 through 5; for participants who will receive only 1 dose of pimodivir on Day 1 [evening], dosing will continue until the morning of Day 6) along with SOC treatment. Participants who meet all treatment extension criteria as defined in the protocol may receive an additional 5 day course of same treatment as received at study start. The SOC treatment is determined by investigator based on local practice, may include influenza antivirals and/or supportive care only. The choice to use influenza antivirals as part of SOC should be started no later than the day when participants initially receive pimodivir. An influenza antiviral as part of SOC cannot be changed (example, switching one influenza antiviral for another) during either treatment period or extension phase, with the exception that an influenza antiviral may be discontinued in case of suspected adverse event (AE).
  Interventions: Drug: Pimodivir 600 mg; Other: SOC Treatment
- Treatment Arm 2 (placebo + SOC treatment) (Placebo Comparator): Participants will receive placebo matching to pimodivir orally twice daily for 5 days (on Days 1 through 5; for participants who will receive only 1 dose of placebo on Day 1 [evening], dosing will continue until morning of Day 6) along with SOC treatment. Participants who meet all treatment extension criteria as defined in protocol may receive an additional 5 day course of same treatment as received at study start. The SOC treatment determined by investigator based on local practice, may include influenza antivirals and/or supportive care only. The choice to use influenza antivirals as part of the SOC should be made before randomization. The influenza antiviral should be started no later than day of first study drug intake. An influenza antiviral as part of the SOC cannot be changed (for example, switching one influenza antiviral for another) during either treatment period/extension phase, with the exception that an influenza antiviral may be discontinued in case of a suspected AE.
  Interventions: Drug: Placebo; Other: SOC Treatment

INTERVENTIONS:
Drug: Pimodivir 600 mg — Participants will receive pimodivir 600 mg orally twice daily for 5 days (on Days 1 through 5; for participants who will receive only 1 dose of pimodivir on Day 1 [evening], dosing will continue until the morning of Day 6). Participants who meet treatment extension criteria may receive an additional 5 day course of the same treatment as received at study start (on Days 6 through 10).
  Arms: Treatment Arm 1 (pimodivir + Standard-of-Care [SOC] treatment)
Drug: Placebo — Participants will receive placebo matching to pimodivir, orally twice daily for 5 days (on Days 1 through 5; for participants who will receive only 1 dose of placebo on Day 1 [evening], dosing will continue until the morning of Day 6). Participants who meet treatment extension criteria may receive an additional 5 day course of the same treatment as received at study start (on Days 6 through 10).
  Arms: Treatment Arm 2 (placebo + SOC treatment)
Other: SOC Treatment — Participants may receive SOC treatment as a part of background therapy. The SOC treatment is determined by the investigator based on local practice, and may include influenza antivirals and/or supportive care only. The choice to use influenza antivirals as part of the SOC should be started no later than the day when participants initially receive pimodivir. An influenza antiviral as part of the SOC cannot be changed (for example, switching one influenza antiviral for another) during either the treatment period or extension phase, with the exception that an influenza antiviral may be discontinued in the case of a suspected AE.

SUMMARY:
The purpose of this study is to evaluate the clinical and virologic benefit of pimodivir in combination with Standard-of-Care (SOC) treatment compared to placebo in combination with SOC treatment.

DETAILED DESCRIPTION:
This double-blind (neither researchers nor participants know what treatment participant is receiving) study will evaluate efficacy/safety of pimodivir in combination with SOC treatment versus placebo in combination with SOC treatment in adolescent, adult, and elderly hospitalized participants with influenza A infection. The study will be conducted in 3 phases: screening phase, double-blind treatment period of 5 days (with the possibility to extend treatment period by 5 days for participants who will enter an optional double-blind extension treatment arm), and post treatment follow-up period of 23 days. Study evaluations will include efficacy, pharmacokinetic, biomarkers, safety and tolerability. The duration of participation in study for each participant is 28 days, except for participants receiving extended treatment, for whom study duration will be up to 33 days.

ELIGIBILITY:
Inclusion Criteria:

* Tested positive for influenza A infection after the onset of symptoms using a polymerase chain reaction (PCR)-based or other rapid molecular diagnostic assay
* Requires hospitalization to treat influenza infection and/or to treat complications of influenza infection (for example, radiological signs of lower respiratory tract disease, septic shock, central nervous system [CNS] involvement, myositis, rhabdomyolysis, acute exacerbation of chronic kidney disease, severe dehydration, myocarditis, pericarditis, ischemic heart disease, exacerbation of underlying chronic pulmonary disease, including asthma, chronic obstructive pulmonary disease [COPD], decompensation of previously controlled diabetes mellitus), including participants admitted to the Intensive Care Unit (ICU)
* Enrollment and initiation of study drug treatment less than or equal to (<=)96 hours after onset of influenza symptoms
* Being on invasive mechanical ventilation or having a peripheral capillary oxygen saturation (SpO2) less than (<)94 percent (%) on room air during screening. Participants with known pre-influenza SpO2 <94% must have an SpO2 decline greater than or equal to (>=)3% from pre-influenza SpO2 during screening
* Having a screening/baseline National Early Warning Score 2 (NEWS2) of >=4

Exclusion Criteria:

* Received more than 3 doses of influenza antiviral medication (for example, oseltamivir [OST] or zanamivir), or any dose of ribavarin (RBV) within 2 weeks, prior to first study drug intake. Received intravenous (IV) peramivir more than one day prior to screening
* Unstable angina pectoris or myocardial infarction within 30 days prior to screening (inclusive)
* Presence of clinically significant heart arrhythmias, uncontrolled, unstable atrial arrhythmia, or sustained ventricular arrhythmia, or risk factors for Torsade de Pointes syndrome
* Known severe hepatic impairment (Child Pugh C cirrhosis) or chronic hepatitis C infection undergoing hepatitis C antiviral therapy
* Severely immunocompromised in the opinion of the investigator (for example, known cluster of differentiation 4 plus [CD4+] count <200 cells per cubic millimeter [cells/mm^3], absolute neutrophil count <750/mm^3, first course of chemotherapy completed within 2 weeks prior to screening, history of stem cell transplant within 1 year prior to screening, any history of a lung transplant)
* Known allergies, hypersensitivity, or intolerance to pimodivir or its excipients

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (268):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Nea Baptist Clinic, Jonesboro, Arkansas
  - UCSF Fresno, Fresno, California
  - Miller Children's at Long Beach Medical Center, Long Beach, California
  - Stanford University School of Medicine, Stanford, California
  - Destin Pulmonary Critical Care, PLLS., Santa Rosa Beach, Florida
  - Northside Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Anne Arundel Medical Center, Annapolis, Maryland
  - University Of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wayne State Univ School of Medicine, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - Western Michigan University Homer Stryker M.D. School of Medicine Center for Clinical Research, Kalamazoo, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital, Troy, Michigan
  - Regents of the University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Saint Michaels Medical Center, Newark, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - Montefiore Medical Center PRIME, The Bronx, New York
  - UC Health LLC, Cincinnati, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Lowcountry Infectious Diseases, Charleston, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - DM Clinical Research, Tomball, Texas
- Argentina (12):
  - Hospital Interzonal General de Agudos Dr. Jose Penna, Bahía Blanca
  - CEMIC (Centro de Educación Médica e Investigaciones Clínicas), C.a.b.a.
  - Hospital Nuestra Señora de la Misericordia, Córdoba
  - Hospital Rawson, Córdoba
  - Hospital San Roque, Córdoba
  - Hospital Cordoba, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Sanatorio Juan XXIII, General Roca
  - Instituto Medico Platense, La Plata
  - Hospital Italiano de La Plata, La Plata Lpl Lpl
  - Hospital Universitario Austral, Pilar
  - Sanatorio Britanico S.A., Rosario
- Australia (6):
  - Flinders Medical Centre, Bedford Park
  - Box Hill Hospital, Box Hill
  - The Alfred Hospital, Melbourne
  - Royal Melbourne Hospital, Melbourne
  - Mater Hospital Brisbane, South Brisbane
  - Townsville Hospital, Townsville
- Austria (3):
  - AKH - Medizinische Universitat Wien, Vienna
  - SMZ Süd - Kaiser Franz Josef Spital Wien, Vienna
  - Social Medizinisches Zentrum Baumgartner Höhe - Otto Wagner Spital, Vienna
- Belgium (3):
  - CHU Saint-Pierre, Brussels
  - Institut Jules Bordet, Brussels
  - ULB Hôpital Erasme, Brussels
- Brazil (11):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Cardresearch - Cardiologia Assistencial, Belo Horizonte
  - Infection Control Ltda, Brasil
  - Associacao Hospitalar Beneficente Sao Vicente de Paulo - Hospital Sao Vicente de Paulo, Passo Fundo
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Irmandade Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Fundacao Jose Luiz Egydio Setubal, São Paulo
  - Hosp. Da Luz Lisboa, São Paulo
- Bulgaria (6):
  - SHATPPD - Ruse Ltd., Rousse
  - SHATPPD - Sofia District EOOD, Sofia
  - Fifth Multiprofile Hospital for Active Treatment - MHAT - Sofia EAD, Sofia
  - Multiprofile Hospital for Active Treatment - MHAT Lyulin EAD, Sofia
  - Military Medical Academy - Sofia, Sofia
  - MHAT Dr Stefan Cherkezov, Veliko Tarnovo
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - Health Sciences North Horizon Sante-Nord, Greater Sudbury, Ontario
- Chile (2):
  - Hospital Dr Sotero del Rio, Puente Alto
  - Hospital El Pino, San Bernardo
- China (4):
  - The Third Xiangya Hospital, Central South University, Changsha
  - Nanfang Hospital, Guangzhou
  - Wuxi People s Hospital, Wuxi
  - Henan Provincial Peoples Hospital, Zhengzhou
- Czechia (3):
  - Fakultni nemocnice Brno, Brno
  - Nemocnice Kyjov, p.o., Kyjov
  - Nemocnice Na Bulovce, Prague
- France (17):
  - Centre Hospitalier d'Agen, Agen
  - CHU Amiens - Hopital Sud, Amiens
  - Hopital Louis Mourier, Colombes
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - CHU Dijon, Dijon
  - Centre Hospitalier Départemental, La Roche S/ Yon Cedex 9
  - CHU de Grenoble Hopital Albert Michallon, La Tronche
  - CHU de Limoges Hopital Dupuytren, Limoges
  - Hopital Edouard Herriot - CHU Lyon, Lyon
  - Hopital Nord Marseille, Marseille
  - CHU Nantes - Hotel Dieu, Nantes
  - CHU De Nice Hopital De l'Archet, Nice
  - Hôpital Bichat - Claude Bernard, Paris
  - Hopital Saint Louis, Paris
  - Hopital Cochin, Paris
  - CHU Poitiers - Hopital la Miletrie, Poitiers
  - CHU Saint Etienne Hopital Nord, Saint-Etienne
- Germany (6):
  - Universitaetsklinikum Koelnt, Cologne
  - Klinikum Donaustauf, Donaustauf
  - Universitaetsklinik Erlangen, Erlangen
  - Universitaetsklinikum Giessen und Marburg GmbH, Hessen
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Klinikum Weiden, Weiden
- Hungary (2):
  - Veszprem Megyei Tudogyogyintezete, Farkasgyepü
  - Tudogyogyintezet Torokbalint, Törökbálint
- India (20):
  - Zydus Hospital-Ahmedabad, Ahmedabad
  - Rajiv Gandhi Institute of Medical Sciences, Balaga
  - M S Ramaiah Memorial Hospital, Bangalore
  - Apollo Hospitals International Limited, Gandhinagar
  - Aware Global Hospital, Hyderabad
  - S. R. Kalla Memorial General Hospital, Jaipur
  - Eternal Heart Care Centre, Jaipur
  - Ajanta Research Cemtre, Lucknow
  - Midland Healthcare & Research Center, Lucknow
  - Vinaya Hospital and Research Center, Mangalore
  - Kasturba Medical College Hospital, Manipal
  - Suretech Hospital and Research Centre Limited, Nagpur
  - Siddhi Hospital, Nashik
  - BLK Super Specialty Hospital, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Fortis Flight Lieutenant Rajan Dhall Hospital, New Delhi
  - Lifepoint Multispecialty Hospital, Pune
  - Sahyadri Speciality Hospital, Pune
  - Shree Giriraj Multispeciality Hospital, Rajkot
  - BAPS Pramukhswami Hospital, Surat
- Israel (14):
  - Haemek Medical Center, Afula
  - Barzilai Medical Center, Ashkelon
  - Soroka University Medical Center, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Campus, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah University Hospita Ein Kerem, Jerusalem
  - Sapir Medical Center, Meir Hospital, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (11):
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico, Milan
  - Fondazione IRCCS Ospedale Maggiore Policlinico,Mangiagalli e Regina Elena, Milan
  - Ospedale San Giuseppe - Fatebenefratelli, Milan
  - Ospedale San Raffaele- Sede Distaccata Ospedale S. Raffaele Turro, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AOU Policlinico di Modena, Modena
  - Azienda Socio Sanitaria Territoriale di Monza Presidio San Gerardo, Monza
  - Azienda Ospedaliera Universitaria Maggiore della Carità, Novara
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Lazzaro Spallanzani IRCCS, Roma
  - Azienda Ospedaliera Universitaria Integrata Verona, Verona
- Latvia (7):
  - Regional Hospital of Liepaja, Liepāja
  - Hospital of Rezekne, Rēzekne
  - Children's Clinical University Hospital, Riga
  - Riga East Clinical University Hospital, Riga
  - Pauls Stradins Clinical University Hospital, Riga
  - Centre of Tuberculosis and Lung Diseases, Riga District
  - Vidzemes Hospital, Valmiera
- Lithuania (3):
  - Klaipeda University Hospital, Klaipėda
  - Siauliai Republican Hospital, Public Institution, Šiauliai
  - Infectious Diseases Center of Vilnius University Hospital Santaros klinikos, Vilnius
- Malaysia (9):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Queen Elizabeth, Kota Kinabalu
  - Hospital Sultanah Nur Zahirah, Kuala
  - Hospital Umum Sarawak, Kuching
  - Hospital Miri, Miri
  - Hospital Tuanku Jaafar, Seremban
  - Hospital Sibu, Sibu
  - Hospital Sungai Buloh, Sungai Buloh
  - Hospital Taiping, Taiping
- Mexico (5):
  - JM Research, SC, Cuernavaca
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Hospital Civil de Guadalajara Dr. Juan I. Menchaca, Guadalajara
  - Hospital Infantil de Mexico Federico Gomez, Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, México
- Netherlands (4):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - UMC Utrecht, Utrecht
  - Gelre Ziekenhuizen Zutphen, Zutphen
- New Zealand (4):
  - Christchurch Hospital, Christchurch
  - Waikato Hospital, Hamilton
  - Tauranga Hospital, Tauranga
  - Wellington Hospital, Wellington
- Clinica Peruano Americana S.A, Trujillo, Peru
- Poland (3):
  - Szpital Miejski ZOZ, Dębica
  - NZOZ Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw
  - Centrum Medyczne w Lancucie Sp.z o.o., Łańcut
- Russia (4):
  - City Hospital #8, Chelyabinsk
  - Clinical Infectious Diseases Hospital n. a. S.P. Botkin, Saint Petersburg
  - LLC Reafarm, Stavropol
  - Clinical Hospital #3, Yaroslavl
- Singapore (3):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Changi General Hospital, Singapore
- Slovakia (4):
  - DFNsP Bratislava, Bratislava
  - Nemocnica Malacky, Nemocnicna A.S., Malacky
  - Nemocnica s poliklinikou S. Kukuru Michalovce, a.s., Michalovce
  - Nemocnica arm. generala L. Svobodu Svidnik, a.s.,, Svidník
- South Africa (8):
  - Clinical Research Centre University of Cape Town, Cape Town
  - Johese Unitas, Centurion
  - Abdullah, IA, Durban
  - Sebastian, Peter, Durban
  - DJW Research, Krugersdorp
  - Emmed Research, Pretoria
  - Into Research, Pretoria
  - Limpopo Clinical Research Initiative, Thabazimbi
- South Korea (13):
  - Chungbuk National University Hospital, Cheongju-si
  - Yonsei University Wonju Severance Christian Hospital, Gangwon-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - The Catholic university of Korea, St. Vincent's Hospital, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Gachon University Gil Medical Center, Incheon
  - The Catholic University of Korea, Incheon St. Mary's Hospital, Incheon
  - Dong-A University Hospital, Pusan
  - Korea University Anam Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
- Spain (17):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Donostia, Donostia / San Sebastian
  - Hosp. Gral. Univ. de Elche, Elche
  - Hosp. Univ. de Getafe, Getafe
  - Hosp. Univ. San Cecilio, Granada
  - Hosp. Univ. Virgen de Las Nieves, Granada
  - Hosp. Univ. de Bellvitge, L'Hospitalet de Llobregat
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Clinico San Carlos, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Hm Monteprincipe, Madrid
  - Hosp. De Mataro, Mataró
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Mutua Terrassa, Terrassa
  - Hosp. Alvaro Cunqueiro, Vigo
- Sweden (3):
  - Department for Heart Failure and Valvular Disease, Malmo
  - Norrlands Universitetssjukhus, Umeå
  - Akademiska Sjukhuset, Uppsala
- Taiwan (4):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Medical University-Wan Fang Hospital, Taipei
- Thailand (4):
  - Siriraj Hospital, Bangkok
  - Bamrasnaradura Infectious Disease Institute, Muang
  - Srinagarind Hospital, Muang
  - Bumrungrad Hospital, Wattana
- Turkey (Türkiye) (6):
  - Hacettepe University Medical Faculty, Ankara
  - Adnan Menderes University, Aydin
  - Dicle University Medical Faculty, Diyarbakır
  - Kocaeli University Medical Faculty, Kocaeli
  - Hacettepe University Medical Faculty, Samanpazarı
  - Karadeniz Teknik University Medical Faculty, Trabzon
- Ukraine (5):
  - Kharkiv MA of PGE Ch of inf.dis. BO Kharkiv Reg.Cl.inf.Hosp., Kharkiv
  - Kyiv Oleksandrivska Clinical Hospital, Kyiv
  - Poltava Regional Clinical Hospital HSEI of Ukraine Ukrainian Medical Stomatological Academy, Poltava
  - CCH #1 Vinnytsia M.I. Pyrogov NMU Ch of Propaedeutics of IM, Vinnytsia
  - Communal Institution Central City Hospital, Zhytomyr
- United Kingdom (5):
  - Aberdeen Royal Infirmary, Aberdeen
  - Western General Hospital, Edinburgh
  - Leeds General Infirmary, Leeds
  - North Manchester General Hospital, Manchester
  - Musgrove Park Hospital, Taunton
- Vietnam (6):
  - Bach Mai Hospital, Hanoi
  - National Hospital for Tropical Diseases, Hanoi
  - Thanh Nhan Hospital, Hanoi
  - Children's Hospital 1, Ho Chi Minh City
  - Children's Hospital 2, Ho Chi Minh City
  - Nguyen Tri Phuong Hospital, Ho Chi Minh City

REFERENCES:
- [Derived] Leopold L, Vingerhoets J, Deleu S, Nalpas C, Weber K, van Dromme I, Lowson D, Michiels B, van Duijnhoven W. Efficacy and Safety of Pimodivir Combined With Standard of Care in Hospitalized and Nonhospitalized High-Risk Adolescents and Adults With Influenza A Infection. J Infect Dis. 2025 Feb 4;231(1):e132-e143. doi: 10.1093/infdis/jiae408. PMID 39172627
- [Derived] Young B, Tan TT, Leo YS. The place for remdesivir in COVID-19 treatment. Lancet Infect Dis. 2021 Jan;21(1):20-21. doi: 10.1016/S1473-3099(20)30911-7. Epub 2020 Nov 26. No abstract available. PMID 33248473

RESULTS

PARTICIPANT FLOW:
Groups:
- Pimodivir + SOC: Participants received 600 milligram (mg) Pimodivir twice daily (bid) on Day 1 through Day 5 along with standard of care (SOC) treatment. Eligible participants were given an optional treatment extension of 5 days bid.
- Placebo + SOC: Participants received matching placebo bid on Day 1 through Day 5 along with SOC treatment. Eligible participants were given an optional treatment extension of 5 days bid.
Period: Overall Study
Arm/Group | Pimodivir + SOC | Placebo + SOC
Started | 168 | 166
Treated | 163 | 163
Completed | 145 | 141
Not Completed | 23 | 25
Not completed — Other | 5 | 1
Not completed — Withdrawal by Subject | 8 | 14
Not completed — Lost to Follow-up | 1 | 7
Not completed — Death | 4 | 0
Not completed — Randomized, not treated | 5 | 3

BASELINE CHARACTERISTICS:
Population: The safety set (or all participants treated) includes all participants who received at least one dose of study drug and were analyzed by treatment arm as treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pimodivir + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 163 | 163 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (15.46) | 57.7 (16.88) | 58.7 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 75 | 167
  Male | 71 | 88 | 159
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 22 | 49
  Not Hispanic or Latino | 132 | 132 | 264
  Unknown or Not Reported | 4 | 9 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 34 | 30 | 64
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 5 | 11 | 16
  White | 113 | 114 | 227
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 3 | 5 | 8
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 4 | 5 | 9
  AUSTRALIA | 1 | 1 | 2
  AUSTRIA | 8 | 10 | 18
  BELGIUM | 0 | 2 | 2
  BRAZIL | 3 | 0 | 3
  BULGARIA | 5 | 5 | 10
  CANADA | 1 | 0 | 1
  CHILE | 0 | 1 | 1
  FRANCE | 2 | 7 | 9
  GERMANY | 0 | 1 | 1
  INDIA | 8 | 10 | 18
  ISRAEL | 20 | 16 | 36
  ITALY | 4 | 0 | 4
  LATVIA | 2 | 1 | 3
  LITHUANIA | 1 | 3 | 4
  MALAYSIA | 12 | 9 | 21
  MEXICO | 7 | 5 | 12
  NETHERLANDS | 1 | 2 | 3
  NEW ZEALAND | 0 | 1 | 1
  POLAND | 12 | 12 | 24
  RUSSIAN FEDERATION | 1 | 0 | 1
  SINGAPORE | 0 | 2 | 2
  SLOVAKIA | 0 | 1 | 1
  SOUTH AFRICA | 9 | 8 | 17
  SPAIN | 13 | 11 | 24
  SWEDEN | 8 | 8 | 16
  TAIWAN | 1 | 0 | 1
  THAILAND | 12 | 10 | 22
  TURKEY | 3 | 5 | 8
  UKRAINE | 6 | 8 | 14
  UNITED KINGDOM | 1 | 0 | 1
  UNITED STATES | 17 | 19 | 36
  VIETNAM | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospital Recovery Scale on Day 6
Description: The hospital recovery scale assesses a participant's clinical status. The scale provides 6 mutually exclusive conditions ordered from best to worst: 1) not hospitalized; 2) non-ICU hospitalization, not requiring supplemental oxygen; 3) non-ICU hospitalization, requiring supplemental oxygen; 4) admitted to the ICU, not requiring invasive mechanical ventilation; 5) requiring invasive mechanical ventilation; and 6) death.
Time Frame: Day 6
Population: Intent-To-Treat infected (ITT-i) set includes all participants from the RAND analysis set who received at least 1 dose of study drug and had a confirmed infection with influenza A. Here, N (number of participants analyzed) defined as participants evaluable for this outcome measure. Here, "n (number analyzed)" is defined as participants analyzed for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 152 | 145
Participants
  Any time since onset influenza: Not hospitalized | 73 | 69
  Any time since onset influenza: Non-ICU hospitalization, not requiring supplemental oxygen | 50 | 42
  Any time since onset influenza: Non-ICU hospitalization, requiring supplemental oxygen | 18 | 25
  Any time since onset influenza: Admitted to the ICU, not requiring invasive mechanical ventilation | 6 | 6
  Any time since onset influenza: Requiring invasive mechanical ventilation | 2 | 3
  Any time since onset influenza: Death | 3 | 0
  Time since onset influenza less than or equal to (<=)72 hour (h): Not hospitalized: number analyzed (Participants) | 122 | 114
  Time since onset influenza less than or equal to (<=)72 hour (h): Not hospitalized | 61 | 56
  Time since onset influenza <=72h: Non-ICU hospitalization, not requiring supplemental oxygen: number analyzed (Participants) | 122 | 114
  Time since onset influenza <=72h: Non-ICU hospitalization, not requiring supplemental oxygen | 38 | 32
  Time since onset influenza <=72h: Non-ICU hospitalization, requiring supplemental oxygen: number analyzed (Participants) | 122 | 114
  Time since onset influenza <=72h: Non-ICU hospitalization, requiring supplemental oxygen | 15 | 19
  Time since onset influenza <=72h: Admitted to the ICU, not requiring invasive mechanical ventilation: number analyzed (Participants) | 122 | 114
  Time since onset influenza <=72h: Admitted to the ICU, not requiring invasive mechanical ventilation | 4 | 5
  Time since onset influenza <=72h: Requiring invasive mechanical ventilation: number analyzed (Participants) | 122 | 114
  Time since onset influenza <=72h: Requiring invasive mechanical ventilation | 2 | 2
  Time since onset influenza <=72h: Death: number analyzed (Participants) | 122 | 114
  Time since onset influenza <=72h: Death | 2 | 0
  Time since onset influenza greater than (>) 72h: Not hospitalized: number analyzed (Participants) | 30 | 31
  Time since onset influenza greater than (>) 72h: Not hospitalized | 12 | 13
  Time since onset influenza >72h: Non-ICU hospitalization, not requiring supplemental oxygen: number analyzed (Participants) | 30 | 31
  Time since onset influenza >72h: Non-ICU hospitalization, not requiring supplemental oxygen | 12 | 10
  Time since onset influenza >72h: Non-ICU hospitalization, requiring supplemental oxygen: number analyzed (Participants) | 30 | 31
  Time since onset influenza >72h: Non-ICU hospitalization, requiring supplemental oxygen | 3 | 6
  Time since onset influenza >72h: Admitted to the ICU, not requiring invasive mechanical ventilation: number analyzed (Participants) | 30 | 31
  Time since onset influenza >72h: Admitted to the ICU, not requiring invasive mechanical ventilation | 2 | 1
  Time since onset influenza >72h: Requiring invasive mechanical ventilation: number analyzed (Participants) | 30 | 31
  Time since onset influenza >72h: Requiring invasive mechanical ventilation | 0 | 1
  Time since onset influenza >72h: Death: number analyzed (Participants) | 30 | 31
  Time since onset influenza >72h: Death | 1 | 0

2. Secondary Outcome: Time to Hospital Discharge
Description: The time to hospital discharge was defined as the time from start of study drug to hospital discharge.
Time Frame: Up to Day 33
Population: The Intent-To-Treat infected (ITT-i) set includes all participants from the RAND (randomized participants with a randomization date time at or before the date time of first intake of study drug, or with a randomization date time and no study drug intake) analysis set who received at least 1 dose of study drug and who had a confirmed infection with influenza A and were analyzed by planned treatment.
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 159 | 159
hours | 113 [94.20 to 118.50] | 108 [92.70 to 116.30]

3. Secondary Outcome: Number of Participants With Adjudicated Influenza Complications
Description: Influenza complications include pulmonary complications (such as respiratory failure, primary viral pneumonia, secondary bacterial pneumonia [including pneumonia attributable to unusual pathogens], exacerbations of chronic underlying pulmonary diseases such as chronic obstructive pulmonary disease [COPD] and asthma) and extrapulmonary complications (such as cardiovascular and cerebrovascular diseases [for example, myocardial infarction, congestive heart failure, arrhythmia, stroke], muscular disorders [for example, myositis, rhabdomyolysis], central nervous system [CNS] involvement, acute exacerbation of chronic kidney disease, decompensation of previously controlled diabetes mellitus, other infections [for example, sinusitis and otitis]).
Time Frame: Up to Day 33
Population: The Intent-To-Treat infected (ITT-i) set includes all participants from the RAND analysis set who received at least 1 dose of study drug and who had a confirmed infection with influenza A and were analyzed by planned treatment. Here, "n (number analyzed)" is defined as number of participants analyzed for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 159 | 159
Participants
  Any time since onset influenza | 28 | 29
  Time since onset influenza <=72h: number analyzed (Participants) | 128 | 126
  Time since onset influenza <=72h | 24 | 24
  Time since onset influenza >72h: number analyzed (Participants) | 31 | 33
  Time since onset influenza >72h | 4 | 5

4. Secondary Outcome: Viral Load Over Time
Description: Viral load over time was measured by quantitative real time polymerase chain reaction (qRT-PCR) and viral culture in the mid-turbinate (MT) nasal swabs and endotracheal samples.
Time Frame: Baseline, Days 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 14 and 19
Population: Intent-To-Treat infected (ITT-i) set includes all participants from the RAND analysis set who received at least 1 dose of study drug and who had a confirmed infection with influenza A. Here, N (number of participants analyzed) defined as participants evaluable for this outcome measure. "n (number analyzed)" is defined as number of participants analyzed for specified category.
Measure: Mean (Standard Deviation); unit: Log 10 viral particles per milliliter
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 153 | 151
Log 10 viral particles per milliliter
  Baseline | 5.657 (1.4693) | 5.655 (1.4117)
  Day 1: number analyzed (Participants) | 3 | 4
  Day 1 | 5.433 (1.3102) | 6.410 (0.7826)
  Day 2: number analyzed (Participants) | 151 | 147
  Day 2 | 4.561 (1.5133) | 4.794 (1.4154)
  Day 3: number analyzed (Participants) | 132 | 125
  Day 3 | 3.913 (1.4202) | 4.057 (1.3425)
  Day 4: number analyzed (Participants) | 109 | 104
  Day 4 | 3.460 (1.4952) | 3.634 (1.2207)
  Day 5: number analyzed (Participants) | 92 | 85
  Day 5 | 3.133 (1.3500) | 3.157 (1.1112)
  Day 6: number analyzed (Participants) | 74 | 68
  Day 6 | 2.552 (0.7100) | 2.876 (0.9750)
  Day 7: number analyzed (Participants) | 4 | 7
  Day 7 | 2.103 (0.0350) | 2.269 (0.3829)
  Day 8: number analyzed (Participants) | 24 | 27
  Day 8 | 2.386 (0.7052) | 2.463 (0.7051)
  Day 9: number analyzed (Participants) | 2 | 7
  Day 9 | 2.050 (0.0000) | 2.611 (0.8281)
  Day 10: number analyzed (Participants) | 138 | 121
  Day 10 | 2.287 (0.6518) | 2.346 (0.6357)
  Day 11: number analyzed (Participants) | 1 | 0
  Day 11 | 2.050 |
  Day 14: number analyzed (Participants) | 135 | 126
  Day 14 | 2.137 (0.4163) | 2.116 (0.2109)
  Day 19: number analyzed (Participants) | 4 | 3
  Day 19 | 2.050 (0.0000) | 2.050 (0.0000)

5. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time Frame: Up to Day 33
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 163 | 163
Participants | 85 | 84

6. Secondary Outcome: Number of Participants With Emergence of Viral Resistance to Pimodivir
Description: Emergence of viral resistance to Pimodivir was detected by genotyping and/or phenotyping. Nasal MT swabs and endotracheal samples were used for sequence analysis of the polymerase basic protein (PB)2 region of the influenza polymerase gene, and of neuraminidase (NA) genes for participants using an NA inhibitor (NAI) as part of their Standard of Care (SOC).
Time Frame: Up to Day 33
Population: Intent-To-Treat infected (ITT-i) set includes all participants from the RAND analysis set who received at least 1 dose of study drug and who had a confirmed infection with influenza A.
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 159 | 159
Participants
  Neuraminidase (NA) region: With emerging mutations of interest | 0 | 3
  Polymerase basic protein (PB) 2 region: With emerging mutations of interest | 2 | 0

7. Secondary Outcome: Plasma Concentration of Pimodivir
Description: Plasma concentration of Pimodivir was reported.
Time Frame: Day 1: 1 hour30minutes to 6 hours postdose, Day 3: Predose, Day 5: Predose and 1 hour30minutes to 6 hours postdose, Day 6: 12 hours postdose
Population: The safety set (or all participants treated) includes all participants who received at least one dose of study drug and were analyzed by treatment arm as treated. Here, N (number of participants analyzed) defined as participants evaluable for this outcome measure. "n (number analyzed)" is defined as number of participants analyzed for specified category.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Pimodivir + SOC
Number analyzed (Participants) | 141
Nanogram per milliliter (ng/mL)
  Day 1: 1 hour30minutes to 6 hours postdose | 1696.3 (2298.4)
  Day 3: Pre-Dose: number analyzed (Participants) | 127
  Day 3: Pre-Dose | 854.3 (898.3)
  Day 5: Pre-Dose: number analyzed (Participants) | 82
  Day 5: Pre-Dose | 940.3 (1081.1)
  Day 5: 1 hour30minutes to 6 hours postdose: number analyzed (Participants) | 79
  Day 5: 1 hour30minutes to 6 hours postdose | 3046.7 (3860.5)
  Day 6: 12hours post dose: number analyzed (Participants) | 55
  Day 6: 12hours post dose | 938.2 (1374.7)

8. Secondary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Tests
Description: Number of participants with clinically significant changes in laboratory tests were reported. Blood samples for hematology, serum chemistry, and urinalysis were collected at predefined time points for clinical laboratory testing.
Time Frame: Up to Day 33
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 163 | 163
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG)
Description: Number of participants with clinically significant changes in Electrocardiogram (ECG) was reported.
Time Frame: Up to Day 33
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 163 | 163
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs
Description: Number of participants with clinically significant changes in vital signs (temperature, pulse rate, respiratory rate and blood pressure) was reported.
Time Frame: Up to Day 33
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Pimodivir + SOC | Placebo + SOC
Number analyzed (Participants) | 163 | 163
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 33
Description: The safety set (or all participants treated) includes all participants who received at least one dose of study drug and were analyzed by treatment arm as treated.
Arm/Group | Pimodivir + SOC | Placebo + SOC
All-Cause Mortality (participants affected / at risk) | 4/163 | 0/163
Serious Adverse Events (participants affected / at risk) | 13/163 | 15/163
Other Adverse Events (participants affected / at risk) | 81/163 | 82/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimodivir + SOC (N=163) | Placebo + SOC (N=163)
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 2 | 0
Cardiac Failure (Cardiac disorders) | 0 | 1
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Pneumonia Bacterial (Infections and infestations) | 0 | 1
Pneumonia Escherichia (Infections and infestations) | 1 | 0
Pneumonia Klebsiella (Infections and infestations) | 0 | 1
Pneumonia Pneumococcal (Infections and infestations) | 0 | 1
Postoperative Wound Infection (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0
Septic Shock (Infections and infestations) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Venous Thrombosis Limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pimodivir + SOC (N=163) | Placebo + SOC (N=163)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Anaemia of Chronic Disease (Blood and lymphatic system disorders) | 0 | 1
Hypereosinophilic Syndrome (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Macrocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 2
Cardiac Failure Acute (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1
Myocardial Ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Dermoid Cyst (Congenital, familial and genetic disorders) | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 2
Cataract (Eye disorders) | 1 | 0
Chalazion (Eye disorders) | 1 | 0
Conjunctivitis Allergic (Eye disorders) | 0 | 1
Dry Eye (Eye disorders) | 1 | 0
Photophobia (Eye disorders) | 1 | 0
Vision Blurred (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 15 | 15
Diarrhoea Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 5
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 7
Oral Pruritus (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Asthenia (General disorders) | 2 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 2 | 1
Malaise (General disorders) | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 1 | 0
Nodule (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 2
Oedema Peripheral (General disorders) | 2 | 3
Peripheral Swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 2
Vessel Puncture Site Bruise (General disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 2
Bronchitis Bacterial (Infections and infestations) | 1 | 0
Candida Infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Clostridium Difficile Colitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Fungal Infection (Infections and infestations) | 1 | 0
Fungal Skin Infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Genital Herpes (Infections and infestations) | 1 | 0
Herpes Simplex (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 1 | 0
Impetigo (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Oral Candidiasis (Infections and infestations) | 2 | 2
Oral Fungal Infection (Infections and infestations) | 1 | 0
Oral Herpes (Infections and infestations) | 2 | 2
Pharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 2
Pneumonia Bacterial (Infections and infestations) | 0 | 1
Pneumonia Haemophilus (Infections and infestations) | 0 | 2
Pneumonia Staphylococcal (Infections and infestations) | 0 | 1
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Septic Shock (Infections and infestations) | 1 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 0 | 1
Superinfection Bacterial (Infections and infestations) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 1
Urinary Tract Infection Staphylococcal (Infections and infestations) | 0 | 1
Vulvovaginal Candidiasis (Infections and infestations) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Haematuria Traumatic (Injury, poisoning and procedural complications) | 1 | 0
Traumatic Haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Alanine Aminotransferase Abnormal (Investigations) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 2
Amylase Increased (Investigations) | 1 | 1
Aspartate Aminotransferase Increased (Investigations) | 1 | 1
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 1
Blood Creatinine Increased (Investigations) | 1 | 0
Blood Uric Acid Increased (Investigations) | 1 | 0
Electrocardiogram Abnormal (Investigations) | 1 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 2
Hepatic Enzyme Increased (Investigations) | 2 | 0
Lipase Increased (Investigations) | 1 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0
Pancreatic Enzymes Increased (Investigations) | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 1
Transaminases Increased (Investigations) | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic Metabolic Decompensation (Metabolism and nutrition disorders) | 1 | 0
Fluid Overload (Metabolism and nutrition disorders) | 1 | 0
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 2
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Ageusia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Dizziness Exertional (Nervous system disorders) | 0 | 1
Dizziness Postural (Nervous system disorders) | 0 | 2
Dysgeusia (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 8 | 8
Intercostal Neuralgia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Psychomotor Hyperactivity (Nervous system disorders) | 1 | 0
Alcohol Withdrawal Syndrome (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Panic Attack (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 1
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypersensitivity Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sputum Increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Macular (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Aortic Dilatation (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 11 | 3
Hypertensive Crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
As the study was terminated early after a pre-planned interim analysis which showed futility, the Sponsor decided not to perform the complete analysis planned per protocol. Hence, data was collected and analyzed for safety and selected efficacy parameters only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT03376321/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03376321/SAP_001.pdf